CLINICAL TRIAL: NCT04144959
Title: STRIDE: A Study of Patients With Lower Extremity Acute Limb Ischemia to Remove Thrombus With the Indigo Aspiration System
Brief Title: A Study of Patients With Lower Extremity Acute Limb Ischemia to Remove Thrombus With the Indigo Aspiration System
Acronym: STRIDE
Status: Completed | Type: Observational
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP 15549
Record Dates: First submitted 2019-10-14; First posted 2019-10-30 (Actual); Results first posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Lower Extremity Acute Limb Ischemia; LE ALI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients with lower extremity acute limb ischemia
  Interventions: Device: Indigo Aspiration System

INTERVENTIONS:
Device: Indigo Aspiration System — Indigo Aspiration System

SUMMARY:
The primary objective of this study is to collect safety and performance data on the Indigo Aspiration System in a patient population with lower extremity acute limb ischemia (LE ALI).

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 18
* Patient presents with acute (≤14 days) occlusion of lower limb artery(ies) (below inguinal ligament)
* Patient with a Rutherford Category I, IIa or IIb score
* Frontline treatment with Indigo Aspiration System
* Informed consent is obtained from either patient or legally authorized representative (LAR)

Exclusion Criteria:

* Life expectancy <1 year
* Vessel size <2 mm
* LE ALI secondary to dissections, vasculitis, and/or target vessel trauma
* Amputation in the ipsilateral limb
* Pregnancy or positive pregnancy test according to site specific standards of care (only required for women of child bearing potential, serum or urine acceptable)
* Absolute contraindication to contrast administration
* Patient is unwilling or unable to comply with protocol follow up schedule and/or based on the Investigator's judgment the patient is not a good study candidate
* Currently participating in an investigational drug or device clinical trial that may confound the study endpoints. Patients in observational, natural history, and/or epidemiological studies not involving intervention are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that present with LE ALI who are eligible for mechanical thrombectomy using the Indigao Aspiration System
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2023-01-02 (Actual); Study Completion 2023-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Maldonado, MD, Principal Investigator — NYU Langone Medical Center
Locations (17):
- United States (14):
  - Stanford University Medical Center, Stanford, California
  - Danbury Hospital, Danbury, Connecticut
  - Manatee Memorial Hospital, Bradenton, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - University of Maryland, Baltimore, Maryland
  - Albany Medical Center, Albany, New York
  - Tisch Hospital NYU Langone Health, New York, New York
  - NC Heart and Vascular Research, Cary, North Carolina
  - Sanger Heart & Vascular Institute, Charlotte, North Carolina
  - Trihealth Good Samaritan Hospital of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Holston Valley Medical, Kingsport, Tennessee
  - Baylor College of Medicine (St. Luke's Medical Center), Houston, Texas
  - Sentara Vascular Specialists, Norfolk, Virginia
- Germany (2):
  - Klinikum rechts der Isar, München
  - St. Franziskus-Hospital - Münster, Münster
- Hospital Clínico Universitario de Santiago, Santiago de Compostela, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maldonado TS, Powell A, Wendorff H, Rowse J, Nagarsheth KH, Dexter DJ, Dietzek AM, Muck PE, Arko FR, Chung J; STRIDE study group. Safety and efficacy of mechanical aspiration thrombectomy for patients with acute lower extremity ischemia. J Vasc Surg. 2024 Mar;79(3):584-592.e5. doi: 10.1016/j.jvs.2023.10.062. Epub 2023 Nov 4. PMID 37931885

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With Lower Extremity Acute Limb Ischemia
Started | 119
Completed | 100 (Completed includes participants who died during follow up.)
Not Completed | 19

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Lower Extremity Acute Limb Ischemia
Number analyzed (Participants) | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 54
  >=65 years | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.3 (13.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 91
  Unknown or Not Reported | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 24
  White | 80
  More than one race | 3
  Unknown or Not Reported | 11

OUTCOME MEASURES:

1. Primary Outcome: Target Limb Salvage Rate
Description: Proportion of participants who did not have a major amputation (above the level of the tarsometatarsal joint)
Time Frame: 1-Month Post Procedure
Population: The analysis population (ITT) contains 111 evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Lower Extremity Acute Limb Ischemia
Number analyzed (Participants) | 111
Participants | 109

2. Secondary Outcome: Technical Success
Description: Defined as TIMI 2/3 flow rate
  TIMI flow grade:
  Grade 0 No perfusion Grade 1 Perfusion past initial occlusion but no distal branch filling. Grade 2 Perfusion with incomplete or slow distal branch filling. Grade 3 Full perfusion with filling of all distal branches.
Time Frame: Immediate Post Procedure
Population: The analysis population (ITT) contains 109 evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Lower Extremity Acute Limb Ischemia
Number analyzed (Participants) | 109
Participants | 105

3. Secondary Outcome: Modified Society for Vascular Surgery Runoff Score
Description: Endpoint is change in modified SVS Runoff Score at post-procedure
  Modified SVS runoff score ranges from 1-19, with a higher score indicating more severe disease
Time Frame: Pre Procedure and immediately Post Procedure
Population: The analysis population (ITT) contains 106 evaluable participants.
Measure: Mean (Standard Deviation); unit: Change in Modified SVS runoff score
Arm/Group | Patients With Lower Extremity Acute Limb Ischemia
Number analyzed (Participants) | 106
Change in Modified SVS runoff score | 6.3 (5.49)

4. Secondary Outcome: Improvement of Rutherford Classification
Description: Improvement of one or more as compared to pre-procedure
  Rutherford classification:
  I.Viable Not immediately threatened
  IIa.Threatened Marginally Salvageable if promptly treated
  IIb. Threatened Immediately Salvageable with immediate revascularization
  III. Irreversible
Time Frame: Up to discharge or 7 days, whichever occurred first
Population: The analysis population (ITT) contains 96 evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Lower Extremity Acute Limb Ischemia
Number analyzed (Participants) | 96
Participants | 83

5. Secondary Outcome: Vessel Patency
Description: Patency is defined as a target lesion without a hemodynamically significant stenosis /reocclusion on duplex ultrasound (>50 %, ) and without target lesion reintervention (TLR ).
Time Frame: 1-Month Post-Procedure
Population: The analysis population (ITT) contains 113 evaluable participants
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Lower Extremity Acute Limb Ischemia
Number analyzed (Participants) | 113
Participants | 101

6. Secondary Outcome: Target Limb Salvage Rate
Description: Proportion of participants who did not have a major amputation (above the level of the tarsometatarsal joint)
Time Frame: 12-Months Post Procedure
Population: The analysis population (ITT) contains 81 evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Lower Extremity Acute Limb Ischemia
Number analyzed (Participants) | 81
Participants | 72

7. Secondary Outcome: Rates of Device Related Serious Adverse Events (SAEs)
Description: A SAE is an event that led to death, led to a serious deterioration in the health of the patient that resulted in life-threatening illness or injury, resulted in chronic disease, resulted in permanent impairment of a body structure or a body function, required in-patient hospitalization or prolongation of existing hospitalization, resulted in medical or surgical intervention to arrest permanent impairment to body structure or a body function, led to fetal distress, fetal death or a congenital abnormality or birth defect
Time Frame: Up until study completion, at approximately 12-Months
Population: The analysis population (ITT) contains 119 evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Lower Extremity Acute Limb Ischemia
Number analyzed (Participants) | 119
Participants | 1

8. Secondary Outcome: Major Bleeding Peri-procedure
Description: Fatal or leading to a drop in hemoglobin of ≥5 g /dl, or significant hypotension with the need for inotropes, or requiring surgery (other than vascular site repair ), or symptomatic intracranial hemorrhage (ICH ), or requiring transfusion of two or three units of red blood cells or equivalent whole blood
Time Frame: within 2 days of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Lower Extremity Acute Limb Ischemia
Number analyzed (Participants) | 119
Participants | 5

9. Secondary Outcome: Mortality
Description: Death due to any cause
Time Frame: 12-Months
Population: The analysis population contains all participants who were enrolled. All deaths within 365 days are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Lower Extremity Acute Limb Ischemia
Number analyzed (Participants) | 119
Participants | 12

ADVERSE EVENTS:
Time Frame: All adverse events are reported for the duration a participant is in the study. All deaths within 365 days are included.
Arm/Group | Patients With Lower Extremity Acute Limb Ischemia
All-Cause Mortality (participants affected / at risk) | 12/119
Serious Adverse Events (participants affected / at risk) | 90/119
Other Adverse Events (participants affected / at risk) | 15/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Lower Extremity Acute Limb Ischemia (N=119)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 5 (5)
Cardiac arrest (Cardiac disorders) | 3 (3)
Cardiac failure (Cardiac disorders) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 3 (3)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Amputation stump pain (General disorders) | 1 (1)
Death (General disorders) | 2 (2)
Impaired healing (General disorders) | 2 (2)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Vascular stent occlusion (General disorders) | 2 (2)
Vascular stent stenosis (General disorders) | 1 (1)
Vascular stent thrombosis (General disorders) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 3 (3)
Cystitis (Infections and infestations) | 1 (1)
Diabetic foot infection (Infections and infestations) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 3 (4)
Postoperative wound infection (Infections and infestations) | 2 (2)
pyelonephritis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 4 (4)
Septic shock (Infections and infestations) | 1 (1)
Skin graft infection (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 4 (6)
Vascular access site infection (Infections and infestations) | 1 (1)
Vascular graft infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 1 (1)
Arterial bypass stenosis (Injury, poisoning and procedural complications) | 1 (1)
Incision site impaired healing (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 2 (2)
Postoperative wound infection (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (2)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 4 (4)
Acute respiratory failure (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 4 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Plantar facial fibromatosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cutaneous T-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Drug withdrawal convulsions (Nervous system disorders) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1)
Generalised tonic clonic seizure (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Multiple sclerosis relapse (Nervous system disorders) | 1 (2)
Seizure (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Mental status change (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Calculus bladder (Renal and urinary disorders) | 1 (1)
Hydroponephrosis (Renal and urinary disorders) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cellulitis (Skin and subcutaneous tissue disorders) | 2 (2)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 1 (1)
Toe amputation (Surgical and medical procedures) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1)
Arterial bypass stenosis (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Haematoma (Vascular disorders) | 2 (2)
Haemorrhage (Vascular disorders) | 16 (16)
Hypertensive urgency (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 2 (2)
Peripheral artery occlusion (Vascular disorders) | 6 (8)
Peripheral artery stenosis (Vascular disorders) | 3 (3)
Peripheral artery thrombosis (Vascular disorders) | 6 (7)
Peripheral embolism (Vascular disorders) | 4 (5)
Peripheral ischaemia (Vascular disorders) | 16 (18)
Vascular dissection (Vascular disorders) | 2 (2)
Vascular pseudoaneurysm (Vascular disorders) | 1 (1)
Vascular stent occlusion (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Lower Extremity Acute Limb Ischemia (N=119)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Postoperative wound infection (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site pain (Injury, poisoning and procedural complications) | 2 (2)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Arterial spasm (Vascular disorders) | 1 (1)
Arterial thrombosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 6 (8)
Peripheral artery occlusion (Vascular disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1)
Vasospasm (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/59/NCT04144959/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-26): https://cdn.clinicaltrials.gov/large-docs/59/NCT04144959/SAP_001.pdf